CLINICAL TRIAL: NCT00520988
Title: Improving Blood Pressure in Colorado
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); Denver Health Medical Center (Other); Colorado Health Outcomes Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCPD08FLA00228
Record Dates: First submitted 2007-08-23; First posted 2007-08-27 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Hypertension
Keywords: hypertension; intervention; disease management; telephone-based; Hypertension: diagnosed but uncontrolled
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Usual care plus use of Interactive Voice Recognition system
  Interventions: Behavioral: Use of telephone-based Interactive Voice Recognition system
- 2 (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Use of telephone-based Interactive Voice Recognition system — Use of telephone-based Interactive Voice Recognition system, for reporting of health information and blood pressure measurements
  Arms: 1

SUMMARY:
We will improve hypertension control in Colorado by implementing a population-based intervention using interactive voice response (IVR) technology that will be delivered to patients in three healthcare systems across Colorado (Denver Health and Hospitals [DH], VA Colorado Healthcare System [VA], and Kaiser Permanente of Colorado [KPCO]). Together, these organizations serve over 1 million Coloradans. The IVR-based hypertension program will: 1) reach out to more patients using fewer resources than a traditional patient visit approach, 2) implement evidence based guidelines for therapy, 3) facilitate patients' acquisition of medications by allowing them to order and receive medications at home, and 4) enhance medication adherence using tailored educational and motivational messages.

HYPOTHESES:

1. A sizable population of patients is at high risk for further cardiovascular morbidity and mortality, based on uncontrolled hypertension.
2. An IVR-centered intervention among patients with diagnosed but uncontrolled hypertension is feasible.
3. An IVR-centered intervention plus usual care for these patients improves BP control, compared to usual care alone.

DETAILED DESCRIPTION:
Hypertension, or high blood pressure (BP), affects 65 million people or almost 1 out of every 4 adults in the U.S. Individuals who have normal BP at 55 years of age have a 90% lifetime risk for developing hypertension. The level of BP elevation is directly related to a person's subsequent risk for heart attack, heart failure, stroke, and kidney failure. In 2002, hypertension was the primary or contributing cause of death in 11% of US deaths and the cost of hypertension was estimated at $59.7 billion. The prevalence of sequelae of uncontrolled hypertension will increase as our population ages unless we develop better programs to control high BP. Hypertension is treatable. If you reduce a person's elevated BP, you reduce their risk of stroke by 30%, heart attack and others forms of coronary heart disease by 20%, congestive heart failure by 50%, and premature death by 10%.3 Despite the evidence supporting hypertension treatment, more than half of patients with hypertension have inadequate BP control.

We will improve hypertension control in Colorado by implementing a population-based intervention using interactive voice response (IVR) technology that will be delivered to patients in three healthcare systems across Colorado (Denver Health and Hospitals [DH], VA Colorado Healthcare System [VA], and Kaiser Permanente of Colorado [KPCO]). Together, these organizations serve over 1 million Coloradans. The IVR-based hypertension program will: 1) reach out to more patients using fewer resources than a traditional patient visit approach, 2) implement evidence based guidelines for therapy, 3) facilitate patients' acquisition of medications by allowing them to order and receive medications at home, and 4) enhance medication adherence using tailored educational and motivational messages. This program will not duplicate or supplant funding for existing programs, but will complement the existing programs which are based on traditional provider-patient encounters.

IVR is a computer-based telephone system that initiates outbound calls, receives inbound calls, and provides information and collects data from patients between office visits. An IVR system has three components: 1) a standard microcomputer, 2) hardware that interfaces with the telephone system to place calls, and 3) software that controls calling operations. Patients require only a telephone to participate in an IVR program. Over 95% of Coloradans have telephones. People are familiar with IVR applications such as systems used by airlines to provide flight information and by healthcare organizations to arrange clinic appointments and refill prescriptions.

*Detailed description of study procedures (duration, description of intervention, study measures, endpoints, specific aims, etc):

Study Visits (both study arms):

At the baseline visit for both study arms, baseline BP will be recorded and patients will be provided educational material. In addition, baseline questionnaires will be completed which includes surveys on medication adherence. Participants assigned to both arms will return to the clinic for a 6 month visit. Prior to the 6 month study visit, all enrolled patients will receive a reminder letter informing them of their pending study appointment. During the 6 month visit, project staff will review the follow up survey, obtain a 6 month blood pressure measurement, assess all current medications, and administer a satisfaction survey.

Usual Care plus IVR arm:

For patients randomized to the usual care plus IVR arm, clinically validated electronic BP cuffs will be provided at no cost to those who do not own one. For patients who own a cuff, they will be asked to bring their cuff to the baseline visit and it will be evaluated by the study staff to determine if it is accurate enough to be used. Patients will be taught the proper technique for using the BP cuffs and will be oriented to the IVR technology and functions. Participants assigned to the usual care plus IVR arm will also meet with the clinical pharmacist to review and adjust as necessary their current medication plan, and establish rapport for the program.

All usual care plus IVR patients will be asked to return at 1 month post-baseline visit, for a blood pressure check, to receive their first blood pressure report in person, and to review the IVR system with study staff if necessary. If medication changes were made at baseline, patients may also need to meet briefly with the clinical pharmacist at the one month visit. If additional clinical pharmacist visits are required beyond the one month visit for laboratory tests or other monitoring of drug changes, these will be provided per current KPCO usual care.

During the 6 months of follow-up, patients in the usual care plus IVR arm will be asked to call in to the IVR system weekly and enter BP measurements from the past week using the touch tone pad on their phone. Through the IVR system, patients will be encouraged to report any symptoms that they have experienced and to ask questions or raise concerns. They can also listen to brief modules on diet, exercise, and smoking cessation. The duration of the call will depend on the number of blood pressure measurements they have to enter and the patient's response to questions. Per JNC VII guidelines, patients will be encouraged to enter a minimum of 4 measurements per week. From previous focus group testing, these calls are expected to take no more than 5-10 minutes. To maximize safety, patients will be instructed to seek immediate medical attention for acute problems, i.e., chest pain and/or if the entered BP measurements exceed a threshold (e.g. SBP>200 mm Hg or DBP>100 mm Hg). An IVR report summarizing the information gathered from the call will be produced and reviewed by a clinical pharmacist. The clinical pharmacist will contact patients if problems are identified or at the patients' request. Based on the BP data provided by the patient, the clinical pharmacist, with physician oversight, will adjust antihypertensive medications or suggest additional medications using national JNC VII hypertension guidelines. This recommendation will be copied to the patient's primary care provider (PCP), along with the IVR BP data. Currently, this system of multidisciplinary management of chronic illness is in place at all three institutions and is accepted by clinicians. Therefore, the management of BP by a clinical pharmacist with physician supervision for the IVR intervention is consistent with usual care at all three sites.

Patients in the usual care plus IVR arm will be instructed to call in weekly to the IVR system for 6 months. During this time, participants will also receive monthly feedback reports in the form of a cover letter and graph of their weekly average blood pressures from their baseline visit through the current month.

At the end of the 6 month study period, if a patient's BP has stabilized at a normal level according to established guidelines, they will "graduate" from the study. Based on prior experience, we expect patients to attain controlled blood pressure in 2-3 months on average, recognizing that some patients will do so more quickly and others more slowly. Therefore, at the end of the 6 month study wave, most of the patients should graduate from the study.

After graduating from the study, patients may continue to enter blood pressure measurements into the IVR system, but the frequency of the calls will not be monitored or enforced. After graduating, patients will still be able to report concerns and ask questions of the clinical pharmacist. For patients who have not reached control by the end of their 6 month visit, they will be referred back to their PCP for BP management and their PCP will be notified of the continued uncontrolled readings.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* have diagnosed but uncontrolled hypertension
* Most recent measurement and one other measurement of the 3 most recent blood pressure measurements in the past 2 years have a systolic pressure >140mmHg or a diastolic pressure >90mmHg. For patients with a diagnosis of diabetes or chronic kidney disease the blood pressure cut-offs will be systolic >130 mm Hg or a diastolic pressure > 80 mm Hg
* not on organizational "do not call" lists or deceased lists
* have been approved for invitation into the study by their physician
* do not have a life-threatening illness
* are not on more than 4 antihypertensive medications
* can use a telephone
* speak either English or Spanish

Exclusion Criteria:

* on organizational "Do Not Call" list or deceased list
* physician does not give permission for them to be included in the study
* younger than 18 years of age
* has a life-threatening illness
* currently takes more than 4 anti-hypertension medications
* does not have or cannot use a phone
* does not speak English or Spanish (languages available in IVR)
* does not want to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2006-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
We will assess the primary measures of effectiveness (control of blood pressure) in the clinic at baseline and 6 months, for both the usual care plus IVR arm and usual care arm alone. | 6 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ho, MD PhD, Principal Investigator — Denver VA Medical Center; Edward Havranek, MD, Principal Investigator — Denver Health Medical Center; David Magid, MD MPH, Principal Investigator — Kaiser Permanente
Locations (3):
- United States (3):
  - Denver Health Medical Center, Denver, Colorado
  - Denver VA Medical Center, Denver, Colorado
  - Kaiser Permanente Colorado, Metro Denver Area, Colorado

REFERENCES:
- [Derived] Welch LK, Olson KL, Snow KE, Pointer L, Lambert-Kerzner A, Havranek EP, Magid DJ, Ho PM. Systolic blood pressure control after participation in a hypertension intervention study. Am J Manag Care. 2011;17(7):473-8. PMID 21819167